CLINICAL TRIAL: NCT05829941
Title: Technology Assisted Treatment for Binge Eating Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HabitAware Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 132180
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HabitAware condition (Experimental): This group will receive the device which messages the participant after a passively detected binge-eating episode with CBT strategies.
  Interventions: Behavioral: Smartwatch app to deliver binge-eating CBT strategies
- Reminder Condition (Placebo Comparator): This group will receive a device that vibrates randomly throughout the day as a reminder not to binge eat.
  Interventions: Behavioral: Reminder control condition

INTERVENTIONS:
Behavioral: Smartwatch app to deliver binge-eating CBT strategies — Participants will receive a smartwatch with a pre-loaded app that will alert the participant to relevant binge-eating strategies based on their previous detected behavior.
  Arms: HabitAware condition
Behavioral: Reminder control condition — Participants will receive a smartwatch that vibrates randomly, and will be instructed the vibration is a cue not to binge eat.
  Arms: Reminder Condition

SUMMARY:
Binge-eating behavior is a central feature of eating disorders (e.g., binge-eating disorder, bulimia nervosa, anorexia nervosa-binge-eating/purging subtype) and is associated with higher rates of psychopathology, psychosocial impairment, medical comorbidity, and more severe obesity, all of which pose significant public health problems. Passive detection of binge eating episodes combined with a context-based reminder intervention could assist a patient in resuming healthy eating patterns. This study will test a smartwatch app that identifies binge eating behavior and provides CBT strategies to the patient after the episode.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. EDE diagnosis of bulimia nervosa or binge eating disorder, with binge-eating episodes occurring at least 2x/week

Exclusion Criteria:

1. Pregnancy or lactation
2. Acute medical or psychiatric risk
3. Psychosis or bipolar disorder (lifetime history)
4. Current substance use disorder within the past six months
5. BMI less than 18.5 kg/m2
6. Acute suicidality requiring hospitalization
7. Food allergies
8. Receiving current psychotherapy
9. On psychotropic medications that have not been on a stable dose for at least six weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in the HabitAware condition that report the treatment is acceptable. | 8 weeks
  Measured via post-treatment survey

SECONDARY OUTCOMES:
Percentage of patients report that the binge episode detection is accurate | 8 weeks
  Measured via post-treatment survey